CLINICAL TRIAL: NCT07277179
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetic Profile and Immunogenicity of Subcutaneous Netakimab in Chinese Adult Patients With Active Ankylosing Spondylitis
Brief Title: Evaluate the Efficacy, Safety, and Pharmacokinetic Profile and Immunogenicity of Subcutaneous Netakimab in Chinese Adult Patients With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SPH-BIOCAD (HK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-085-CN02
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — netakimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Netakimab (Experimental): Netakimab administered by subcutaneous injection until Week 52
  Interventions: Drug: Netakimab
- Placebo (Placebo Comparator): Placebo administered by subcutaneous injection until Week 16 then Netakimab subcutaneous injection until 52 week
  Interventions: Drug: Netakimab; Drug: Placebo

INTERVENTIONS:
Drug: Netakimab — Netakimab administered subcutaneously
Drug: Placebo — Placebo administered subcutaneously
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to To evaluate the efficacy of subcutaneous (SC) Netakimab in adult Chinese patients with Active Ankylosing Spondylitis. Researchers will compare Netakimab to placebo to see if Netakimab works to treat Ankylosing Spondylitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients fully understand the objectives, procedures and possible adverse reactions of this study, voluntarily participate in the study and sign the informed consent form (ICF) approved by the Institutional Ethics Committee (IEC).
2. Male or female aged 18-65 years (inclusive) on the day of signing the ICF.
3. Patients meet the diagnostic criteria for ankylosing spondylitis (New York criteria as modified in 1984) and have a history of back pain for ≥ 3 months, with onset age < 45 years.
4. BASDAI score ≥ 4 at screening and baseline, and a spinal pain score [using a 0-10-point numerical rating scale (NRS)] of ≥ 4.
5. Suboptimal or no response to NSAIDs.
6. For patients taking NSAIDs regularly as treatment for ankylosing spondylitis, a stable dose of at least 2 weeks is required to be maintained prior to randomization.
7. At screening, if patients have received or are receiving a TNF-α inhibitor (not more than 1), the duration of administration must be no less than 3 months (at an approved dose) and the patients have a poor efficacy or are intolerant of the TNF-α inhibitor.
8. Female patients should have a negative blood pregnancy test.

Exclusion Criteria:

1. Complete ankylosis of spine joint with syndesmophyte on the cervical vertebra, thoracic vertebra, and lumbar vertebra sides of all intervertebral spaces.
2. Patients who are known to be allergic to any component of the investigational product or other excipients.
3. Prior use of any monoclonal antibody targeting interleukin 17 (IL-17) or interleukin 17 receptor (IL-17R), IL-12/23, or any other monoclonal antibodies for the treatment of ankylosing spondylitis (except for antibodies targeting TNFα)
4. Current or previous tuberculosis (TB) infection or latent TB
5. History of lymphoproliferative disorders such as lymphoma, or current signs and symptoms suggestive of lymphoproliferative disorders.
6. Any active malignancy or history of malignancy (with the exception of squamous carcinoma in situ or basal cell carcinoma of the skin or cervical cancer in situ with curative outcome) within 5 years prior to screening.
7. Major surgery (including joint surgery) within 3 months prior to screening, or surgery planned during the study.
8. Patients who have the following active infections or history of infections:
9. Presence of hepatitis B [hepatitis B surface antigen positive (HBsAg +), or anti-hepatitis B core antibody positive (HBcAb +) and HBV DNA positive], hepatitis C [hepatitis C antibody (anti-HCV Ab) positive and HCV-RNA positive], human immunodeficiency virus (HIV), or syphilis infection.
10. A history of epileptic seizure or convulsion.
11. Chronic intestinal inflammatory disease (except 'rohn's disease, nonspecific ulcerative colitis).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving ASAS40 | Week 16
  Proportion of patients achieving 40% improvement criteria established by the International Ankylosing Spondylitis Assessment Task Force at Week 16.

SECONDARY OUTCOMES:
Proportion of patients achieving ASAS20 | at Week 2, 4, 8, 12, 16, 24, 36, and 52.
  Proportion of patients achieving 20% improvement criteria established by the International Ankylosing Spondylitis Assessment Task Force at Week 2, 4, 8, 12, 16, 24, 36, and 52.
Proportion of patients achieving ASAS40 | at Week 2, 4, 8, 12, 24, 36, and 52
  Proportion of patients achieving 40% improvement criteria established by the International Ankylosing Spondylitis Assessment Task Force at Week 2, 4, 8, 12, 24, 36, and 52.
Proportion of patients achieving ASAS5/6 | at Week 2, 4, 8, 12, 16, 24, 36, and 52
  Proportion of patients achieving ASAS5/6 at Week 2, 4, 8, 12, 16, 24, 36, and 52.
Change from baseline in BASDAI | at Week 2, 4, 8, 12, 16, 24, 36, and 52.
  Change from baseline in BASDAI at Week 2, 4, 8, 12, 16, 24, 36, and 52.
Change from baseline in BASMI | at Week 2, 4, 8, 12, 16, 24, 36, and 52
  Change from baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 2, 4, 8, 12, 16, 24, 36, and 52
Change from baseline in BASFI | at Week 2, 4, 8, 12, 16, 24, 36, and 52
  Change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 2, 4, 8, 12, 16, 24, 36, and 52.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No